CLINICAL TRIAL: NCT03745118
Title: Development of a Practical, Minimally Invasive Seizure Gauge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Benjamin H. Brinkmann, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-008357
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy
Keywords: Seizure
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Monitoring Device (Other): Subjects will be asked to wear up to 4 different noninvasive seizure detection devices including EpiTel EpiLog, Byte Flies Sensor Dots, Empatica E4, Biovotion Everion, GeneActiv
  Interventions: Device: EpiTel EpiLog; Device: Byte Flies Sensor Dots; Device: Empatica E4; Device: Biovotion Everion; Device: GeneActiv

INTERVENTIONS:
Device: EpiTel EpiLog — Plastic pad that is about the size of a house key, and will be adhered to your scalp with gel
  Other Names: Epilog
Device: Byte Flies Sensor Dots — Plastic pads that will be adhered to your chest area
  Other Names: Byteflies; Sensor Dots
Device: Empatica E4 — wearable seizure detection wristband
  Other Names: E4 Wristband
Device: Biovotion Everion — wearable seizure detection device armband that is attached to upper arm
Device: GeneActiv — wearable seizure detection watch

SUMMARY:
The researchers are trying to assess changes in physiological signals before and during seizures.

DETAILED DESCRIPTION:
Subjects that are undergoing video EEG monitoring in the hospital for their epilepsy at Mayo Clinic will be consented to participate in this study for a minimum of two days and/or the duration of their hospital stay for their clinical care. Subjects will be asked to wear up to 4 different commercially available seizure detection devices and complete surveys.

In the second year of the study patients who have implanted devices capable of recording or detecting seizures will be recruited to wear a noninvasive biosensor for multiple months. This data will be used to develop algorithms capable of detecting and/or forecasting seizures.

When the subjects clinical EEG monitoring is completed data scientists will analyze the data to identify patterns.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epilepsy- scalp EEG or invasive EEG monitoring for clinical care, or an implanted device capable of monitoring brain activity and identifying seizures (e.g. NeuroPace RNS, Medtronic PC+S, Medtronic RC+S)
* Pediatric subjects 7 years of age or older.

Exclusion Criteria:

* Cognitive or psychiatric condition rendering patient unable to cooperate with data collection, or manage and recharge smart watch and tablet computer devices.
* Presence of open or healing wounds near monitoring sites (infection risk).

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Assessment of Physiological Signals Measurable with Wearable Sensors | 2-10 days approximately
  We will collect physiological signals with the five wearable, noninvasive biosensors listed below in Mayo patients undergoing scalp-recorded video EEG and invasive stereotactic EEG/video monitoring as part of their clinical epilepsy evaluation. We will evaluate biosignals based on data quality and reliability, and subject comfort and ease of use.
Pattern Analysis | 2-10 days approximately
  We will apply data mining and machine learning methods to search for patterns in the collected physiological signals and correlate these patterns with the timing of seizures identified by the patient's clinical video-EEG monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin (Ben) H. Brinkmann, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials